CLINICAL TRIAL: NCT02997735
Title: Parent eReferral to Tobacco Quitline in Primary Care
Brief Title: Parent eReferral to Tobacco Quitline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 16-012868
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Secondhand Smoke
Keywords: Secondhand Smoke; Nicotine Replacement Therapy; Clinical Decision Support; Tobacco quitline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic Quitline Referral (Experimental): The electronic quitline referral will be embedded within the Tobacco Treatment CDS tool, a CDS system previously developed to help pediatricians provide smoking cessation counseling and treatment to parents who smoke, modeled off the CEASE intervention, an evidence-based approach for implementing smoking cessation treatment of parents in the pediatric setting. The parental tobacco treatment CDS tool prompts the pediatric clinician to ask the parent about smoking status and assess interest in quitting (at all well-child and acute visits), links to an electronic nicotine replacement therapy prescription for parents interested in quitting, and guides appropriate documentation. Electronic referral to the quitline will be made by clicking an automated link embedded in the tool that will send the parent smokers' names and telephone numbers (entered by the clinician) directly to the Pennsylvania (PA) Free Quitline.
  Interventions: Behavioral: Quitline Delivered Treatment
- Standard of Practice (Other): All procedures implemented in the standard referral approach will be identical to those in the electronic referral approach with the exception of providing the telephone number for the Quitline to the parent (rather than electronic referral). The clinician workflow will be nearly the same, in that the clinician will use the link embedded in the tobacco treatment CDS tool to add the quitline to the patient's discharge paperwork (rather than automatically refer to the quitline).
  Interventions: Behavioral: Quitline Delivered Treatment

INTERVENTIONS:
Behavioral: Quitline Delivered Treatment — The PA Free quitline is funded by the Pennsylvania Department of Health and staffed by trained cessation counselors available 24 hours a day, 7 days a week. Counseling is available in English and Spanish and can be provided in at least 15 additional languages through a third party. All smokers who enroll in smoking cessation treatment will receive counseling and support consistent with accepted clinical practice guidelines. This treatment includes as many as 5 proactive counseling calls, each designed to help develop problem-solving and coping skills, secure social support, and plan for long-term abstinence. Participants can also call an 800 telephone number as needed for additional support between calls. The timing of counseling calls will be relapse sensitive and include a call 1-2 days after the quit date, another telephone call a week after the first call, and additional calls generally occurring at 2-3-week intervals thereafter.

SUMMARY:
Secondhand smoke (SHS) exposure is a significant public health problem in that it both harms children and is widely prevalent, affecting more than 40% of US children. Tobacco cessation quitlines are effective in helping smokers quit, but few smokers make use of their services. Electronic health record-based systems that automate referral of interested parents to quitlines through pediatric settings may increase the proportion of smokers who successfully enroll in treatment.

DETAILED DESCRIPTION:
This is a randomized controlled study of electronic quitline referral compared to standard practice. Parent enrollment in the quitline will be reported to the study team by the state tobacco quitline, managed by the Pennsylvania Department of Health.

This is a single site study at one large outpatient pediatric practice. Eligible study participants are parents/caregivers (hereafter referred to as "parents"), 18 years of age or older, who are present for the child's healthcare (both well-child and acute) visit, who smoke, and who are interested in receiving treatment through the tobacco quitline.

The intervention is electronic referral to the tobacco quitline for parent smokers. The referral process will be embedded in a tobacco treatment clinical decision support (CDS) tool, created to help pediatricians provide counseling and treatment to parent smokers. The primary outcome of interest is smoker enrollment in the quitline, defined as the proportion of parent smokers identified in the clinic that enroll in quitline treatment compared across the intervention (electronic referral) and control (standard practice) approaches. Secondary outcomes include patient and parent demographic and behavioral factors associated with successful enrollment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Parent/caregiver who presents for their child's healthcare (both well-child and acute) visit
* Current smoker
* Interested in being referred to the tobacco quitline

Exclusion Criteria:

* Less than 18 years of age
* Parent/caregiver who smokes but is not present during their child's healthcare visit
* Not interested in referral to the tobacco quitline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2017-01-11; Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenssen BP, Muthu N, Kelly MK, Baca H, Shults J, Grundmeier RW, Fiks AG. Parent eReferral to Tobacco Quitline: A Pragmatic Randomized Trial in Pediatric Primary Care. Am J Prev Med. 2019 Jul;57(1):32-40. doi: 10.1016/j.amepre.2019.03.005. Epub 2019 May 21. PMID 31122792

RESULTS

PARTICIPANT FLOW:
Groups:
- eReferral: Pediatricians screened for tobacco use; smokers were given brief advice to quit and, if interested in quitting, were referred to the quitline. The eReferral ("warm handoff") involved electronically sending parent information to the quitline (parent received a call within 24-48 hours).
- Control: Pediatricians screened for tobacco use; smokers were given brief advice to quit and, if interested in quitting, were referred to the quitline. The eReferral ("warm handoff") involved electronically sending parent information to the quitline (parent received a call within 24-48 hours). Control group procedures were identical to eReferral, except the quitline number was provided to the parent.
Period: Overall Study
Arm/Group | eReferral | Control
Started | 233 | 251
Completed | 233 | 251
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Rows may not add up to total owing to either not reported or missing data.
Groups:
- eReferral: Pediatricians screened for tobacco use; parent smokers were given brief advice to quit and, if interested in quitting, were referred to the quitline. The eReferral ("warm handoff") involved electronically sending parent information to the quitline (parent received a call within 24-48 hours).
- Control: Pediatricians screened for tobacco use; parent smokers were given brief advice to quit and, if interested in quitting, were referred to the quitline. The eReferral ("warm handoff") involved electronically sending parent information to the quitline (parent received a call within 24-48 hours). Control group procedures were identical to eReferral, except the quitline number was provided to the parent.
- Total: Total of all reporting groups
Arm/Group | eReferral | Control | Total
Number analyzed (Participants) | 233 | 251 | 484
Age, Customized [Count of Participants; unit: Participants] — Parent Age
  Participants
    18-24 | 20 | 23 | 43
    25-34 | 107 | 122 | 229
    35-49 | 87 | 82 | 169
    50 or greater | 18 | 21 | 39
    Not available | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Child Sex
  Participants
    Female | 103 | 118 | 221
    Male | 130 | 133 | 263
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Child Ethnicity
  Participants
    Hispanic or Latino | 20 | 8 | 28
    Not Hispanic or Latino | 213 | 240 | 453
    Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Child Race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 3 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 213 | 225 | 438
    White | 5 | 4 | 9
    More than one race | 4 | 2 | 6
    Unknown or Not Reported | 9 | 16 | 25
Child age [Count of Participants; unit: Participants]
  <1 | 43 | 42 | 85
  1-5 | 89 | 82 | 171
  6-12 | 78 | 96 | 174
  13 or older | 23 | 29 | 52
  Not available | 0 | 2 | 2
Insurance status (child) [Count of Participants; unit: Participants]
  Private | 33 | 27 | 60
  Medicaid | 197 | 219 | 416
  Self-pay | 3 | 4 | 7
  Not available | 0 | 1 | 1
Asthma diagnosis (child) [Count of Participants; unit: Participants]
  No asthma | 168 | 176 | 344
  Asthma | 65 | 75 | 140
Cigarettes smoked per day (Parent) [Count of Participants; unit: Participants]
  < 10 | 138 | 165 | 303
  10 or greater | 93 | 82 | 175
  Not available | 2 | 4 | 6
Quit stage (Parent) [Count of Participants; unit: Participants]
  30 days | 124 | 133 | 257
  6 months | 76 | 71 | 147
  Over 6 months | 30 | 41 | 71
  Not Available | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Parent Smokers Who Enrolled in Quitline
Description: Proportion of parent smokers identified in clinic that enroll in quitline treatment compared across the intervention (electronic referral) and control (standard of practice) approaches. Primary analysis wibased on an intent to treat approach and includes all subjects randomized at their referral visit.
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 233 | 251
Participants
  Not Enrolled | 209 | 245
  Enrolled | 24 | 5
  Missing | 0 | 1

2. Secondary Outcome: Number of Calls With the Quitline
Description: Total number of parent contacts with the quitline post-enrollment, compared between intervention and control and reported by the PA Quitline
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 233 | 251
Participants
  No calls | 209 | 245
  One call (enrollment only) | 7 | 0
  Two calls | 12 | 3
  Three or more calls | 5 | 2
  Missing | 0 | 1

3. Secondary Outcome: Number of Parents Who Quit Smoking
Description: Self-reported parent quit rates post-enrollment, compared between the intervention and control and reported by the PA Quitline
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 233 | 251
Participants | 1 | 0

4. Other Pre Specified Outcome: Characteristics Associated With Successful Quitline Enrollment, Study Arm
Description: Multivariable logistic regression was used to assess demographic and behavioral factors which independently associated with successful enrollment. The Odds Ratios (ORs) from multivariable logistic regression model of characteristics associated with successful quitline enrollment.
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 233 | 251
Participants | 24 | 5
Statistical Analysis 1: Comparison: eReferral vs Control; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 7.78, 95% CI 2-sided [2.81 to 27.90] — ORs from multivariable logistic regression model of characteristics associated with successful quitline enrollment

5. Other Pre Specified Outcome: Characteristics Associated With Successful Quitline Enrollment, Patient Age
Description: Multivariable logistic regression was used to assess demographic and behavioral factors which independently associated with successful enrollment.
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 233 | 249
Participants
  <1 | 43 | 42
  1-5 | 89 | 82
  6-12 | 78 | 96
  13 or older | 23 | 29
Statistical Analysis 1: Comparison: eReferral vs Control; Test type: Superiority; p = 0.15, Chi-squared; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.13 to 1.72] — 1-5 years Row (<1 Ref)
Statistical Analysis 2: Comparison: eReferral vs Control; Test type: Superiority; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.18 to 2.12] — 6-12 years Row (<1 Ref)
Statistical Analysis 3: Comparison: eReferral vs Control; Test type: Superiority; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.49 to 6.94] — 13 or Older Row (<1 Ref)

6. Other Pre Specified Outcome: Characteristics Associated With Successful Quitline Enrollment, Parent Age
Description: as for outcome 5
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 232 | 248
Participants
  18-34 | 127 | 145
  35-49 | 87 | 82
  50 or older | 18 | 21
Statistical Analysis 1: Comparison: eReferral vs Control; Test type: Superiority; p = 0.028, Chi-squared; Odds Ratio (OR) = 2.38, 95% CI 2-sided [0.92 to 6.50] — 35-49 years Row (18-34 Ref)
Statistical Analysis 2: Comparison: eReferral vs Control; Test type: Superiority; Odds Ratio (OR) = 5.10, 95% CI 2-sided [1.46 to 17.32] — 50 or older Row (18-34 Ref)

7. Other Pre Specified Outcome: Characteristics Associated With Successful Quitline Enrollment, Asthma Diagnosis (Child)
Description: as for outcome 5
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 233 | 250
Participants
  No asthma | 168 | 176
  Asthma | 65 | 74
Statistical Analysis 1: Comparison: eReferral vs Control; Test type: Superiority; p = 0.85, Chi-squared; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.40 to 2.80] — Asthma Row (No asthma Ref)

8. Other Pre Specified Outcome: Characteristics Associated With Successful Quitline Enrollment, Cigarettes Smoked Per Day
Description: as for outcome 5
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 231 | 247
Participants
  <10 | 138 | 165
  10 or more | 93 | 82
Statistical Analysis 1: Comparison: eReferral vs Control; Test type: Superiority; p = 0.086, Chi-squared; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.90 to 6.50] — 10 or more cigarettes Row (<10 cigarettes Ref)

9. Other Pre Specified Outcome: Characteristics Associated With Successful Quitline Enrollment, Quit Stage
Description: as for outcome 5
Time Frame: Through study completion, up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | eReferral | Control
Number analyzed (Participants) | 230 | 245
Participants
  30 days | 124 | 133
  Less than 6 months | 76 | 71
  6 or more months | 30 | 41
Statistical Analysis 1: Comparison: eReferral vs Control; Test type: Superiority; p = 0.35, Chi-squared; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.15 to 1.27] — Less than 6 months Row (30 days Ref)
Statistical Analysis 2: Comparison: eReferral vs Control; Test type: Superiority; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.15 to 2.21]; 6 or more months Row (30 days Ref)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | eReferral | Control
All-Cause Mortality (participants affected / at risk) | 0/233 | 0/251
Serious Adverse Events (participants affected / at risk) | 0/233 | 0/251
Other Adverse Events (participants affected / at risk) | 0/233 | 0/251

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT02997735/Prot_SAP_000.pdf